CLINICAL TRIAL: NCT00656175
Title: Phase II Study of Raltegravir as Replacement for Protease Inhibitor or Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) Based Antiretroviral Therapy in Women With Fat Accumulation
Brief Title: Raltegravir Therapy for Women With HIV and Fat Accumulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Case Western Reserve University (Other); Vanderbilt University (Other); Tufts University (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Judith S. Currier, M.D., University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IISP-Raltegravir; NCT00755612 (obsolete NCT alias)
Record Dates: First submitted 2008-04-02; First posted 2008-04-10 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: lipodystrophy; fat; visceral fat; HIV; women; raltegravir; ART; anti HIV therapy; NNRTI; Protease inhibitor; integrase inhibitor; treatment experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Platelet Glycoprotein IV Deficiency | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (Active Comparator): Immediate switch of PI or NNRTI to Raltegravir
  Interventions: Drug: raltegravir
- Delayed (Active Comparator): Continue current therapy unchanged for 24 weeks, then switch PI or NNRTI to Raltegravir
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — raltegravir
  Other Names: Isentress

SUMMARY:
Ritonavir-boosted protease inhibitor (PI) regimens have become a backbone for treatment of people with HIV. However, adverse drug effects, particularly lipodystrophy/lipoatrophy are closely associated with these regimens. Therefore, there is a need for a drug with comparable effectiveness to the ritonavir boosted PIs without the side effects of dyslipidemia, which has been associated with elevated cholesterol and cardiovascular disease

Raltegravir is an HIV integrase inhibitor in phase III clinical development. To date there are no approved drugs that target the same stage of the HIV-1 lifecycle. However, data from studies indicate that raltegravir is generally safe and well tolerated and has strong antiretroviral activity when used in combination with licensed antiretroviral medications.

This study aims to demonstrate that patients substituting raltegravir for a PI or NNRTI based antiretroviral regimen will be associated with a 10% reduction in body fat over 24 weeks.

The study will consist of a total of 10 subject visits over a period of 48 weeks. Approximately 40 female patients will participate in this study (approximately 10 at UCLA).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry or plasma HIV-1 RNA > 2000 on two occasions,
* Female subjects 18 years or older
* Documented central fat accumulation (defined by waist circumference of > 94 cm or a waist to hip ratio of > 0.88).
* Documented HIV RNA <50 copies/mL at screening and <400 copies/mL in the past 6 months.
* Current antiretroviral therapy with two nucleoside analogues and either a non-nucleoside analogue (nevirapine, efavirenz or TMC125) or an approved protease inhibitor. Patients on NNRTI+PI at study entry will be excluded. Study participants do not need to be on their first regimen. No changes in ART in the 12 weeks prior to screening. The nucleoside backbone must include either tenofovir or abacavir and either lamivudine or emtricitabine. Fixed dose combinations with emtricitabine or abacavir are allowed.
* For females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy, or bilateral oophorectomy and/or tubal ligation), will need a negative serum or urine pregnancy test within 48 hours prior to entry.
* Ability and willingness of subject to provide informed consent.

Exclusion Criteria:

* Pregnancy: current or within the past 6 months or breast feeding
* Prior treatment history that would preclude the use of emtricitabine or abacavir as the nucleoside backbone during study treatment
* Current use of metformin or thiazolidinediones.
* Use of growth hormone or growth hormone releasing factor in the last 6 months before screening.
* Change or initiation of anti-hyperlipemic regimen within 3 months prior to randomization; Use of stable anti-hyperlipemic regimen during the study is allowed.
* Current use of androgen therapy.
* Intent to modify diet, exercise habits or to enroll in a weight loss intervention during the study period.
* Current or projected need to use rifampin, dilantin or phenobarbital during the 48-week study period.
* Laboratory values at screening of

  * ANC >500 cells/mm3
  * Hemoglobin <10 gm/dl
  * CrCl > 60 ml/min (estimated by Cockcroft-Gault equation)
  * AST or ALT > 3 x ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Currier, M.D., Principal Investigator — University of California, Los Angeles; Grace McComsey, M.D., Study Chair — Case School of Medicine
Locations (5):
- United States (4):
  - UCLA CARE Center, Los Angeles, California
  - Tufts University School of Medicine, Boston, Massachusetts
  - Case School of Medicine, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
- University Health Network, Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lake JE, McComsey GA, Hulgan TM, Wanke CA, Mangili A, Walmsley SL, Boger MS, Turner RR, McCreath HE, Currier JS. A randomized trial of Raltegravir replacement for protease inhibitor or non-nucleoside reverse transcriptase inhibitor in HIV-infected women with lipohypertrophy. AIDS Patient Care STDS. 2012 Sep;26(9):532-40. doi: 10.1089/apc.2012.0135. Epub 2012 Jul 23. PMID 22823027
- [Derived] Offor O, Utay N, Reynoso D, Somasunderam A, Currier J, Lake J. Adiponectin and the steatosis marker Chi3L1 decrease following switch to raltegravir compared to continued PI/NNRTI-based antiretroviral therapy. PLoS One. 2018 May 10;13(5):e0196395. doi: 10.1371/journal.pone.0196395. eCollection 2018. PMID 29746485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 subjects were screened, 39 enrolled, and 37 completed the Week 24 primary endpoint at 5 sites in North America.
  Of the 37 subjects included in the as-treated analysis, 17 were randomized to immediate-switch (Immediate Group), and 20 to delayed-switch (Delayed Group).
Groups:
- Immediate: Immediate switch of PI or NNRTI to Raltegravir (400 mg twice daily)
- Delayed: Continue current therapy unchanged for 24 weeks, then switch PI or NNRTI to Raltegravir (400mg twice daily)
Period: Overall Study
Arm/Group | Immediate | Delayed
Started | 18 | 21
Completed | 17 | 20
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Transportation issues | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Delayed: Continue current therapy unchanged for 24 weeks then switch PI or NNRTI to Raltegravir
- Total: Total of all reporting groups
Arm/Group | Immediate | Delayed | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 39
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (47) | 36 (51) | 37 (49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Subjects were recruited from 5 centers in North America between September 2008 and July 2010. Age 18 or older, documented HIV-1 infection, central fat accumulation at screening and <400 copies/mL for the 6 months prior to entry, current ART with a nucleoside (NRTI) backbone of tenofovir or abacavir AND emtricitabine or lamivudine PLUS either a PI or NNRTI, no change in ART for 12 weeks prior to screening, and ability and willingness to provide informed consent.
  Participants
    African-American | 9 | 13 | 22
    Hispanic | 5 | 3 | 8
    White | 3 | 5 | 8 [lower limit 24]
    Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants] — Subjects were recruited from 5 centers in North America between September 2008 and July 2010.
  Participants
    North America | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Baseline to 24-week Change in Visceral Adipose Tissue Volume (cm^2)
Description: Adipose tissue volumes were measured via single slice L4-L5 CT scan, and volumes were calculated using cm^2, not cm^3, as is standard protocol at the Tufts University Body Composition Reading Center. The authors acknowledge that cm^2 uses area as a surrogate for volume, but this protocol is well-accepted in our field.
Time Frame: Baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 17 | 20
cm^2 | -6.6 [-15.5 to 17.6] | 1.8 [-9.3 to 8.1]
Statistical Analysis 1: Comparison: Immediate vs Delayed; Wilcoxon sign-rank test used for statistical significance; Test type: Superiority or Other; p = 0.52, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Immediate | Delayed
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

LIMITATIONS AND CAVEATS:
High prevalence of generalized obesity; small sample size; short follow-up; not designed to assess the potential contribution of NRTIs to lipohypertrophy, nor could we exclude the NRTI backbone as a confounding factor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes